CLINICAL TRIAL: NCT06292559
Title: A Randomized Prospective Study Between STN-DBS and GPi-DBS in Meige Syndrome
Brief Title: A Comparison Between STN-DBS and GPi-DBS in Meige Syndrome Evaluated by Flexible Electrodes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STN or GPi in Meige Syndrom
Record Dates: First submitted 2024-02-16; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-11

CONDITIONS: Meige Syndrome
Keywords: DBS; STN vs GPi
MeSH Terms: conditions — Meige Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral STN deep brain stimulation (Placebo Comparator): Patients with Meige syndrome accepted STN DBS
  Interventions: Device: Bilateral STN deep brain stimulation
- Bilateral GPi deep brain stimulation (Experimental): Patients with Meige syndrome accepted GPi DBS
  Interventions: Device: Bilateral GPi deep brain stimulation

INTERVENTIONS:
Device: Bilateral STN deep brain stimulation — patients with Meige syndrome underwent bilateral subthalamic stimulation
  Arms: Bilateral STN deep brain stimulation
Device: Bilateral GPi deep brain stimulation — patients with Meige syndrome underwent bilateral pallidal stimulation
  Arms: Bilateral GPi deep brain stimulation

SUMMARY:
Deep-brain stimulation (DBS) is an effective treatment for patients with Meige syndrome. The globus pallidus interna (GPi) and the subthalamic nucleus (STN) are both accepted targets for this treatment. Researchers designed this study to compare the 12-month outcomes for patients who undergo bilateral stimulation of the GPi or STN.

DETAILED DESCRIPTION:
Deep-brain stimulation (DBS) is an effective treatment for patients with Meige syndrome. The globus pallidus interna (GPi) and the subthalamic nucleus (STN) are accepted targets for this treatment. Researchers are willing to compared12-month outcomes for patients who had undergone bilateral stimulation of the GPi or STN. Forty-two Asian patients with primary Meige syndrome who underwent GPi or STN neurostimulation were recruited between Nov. 2023 and Nov. 2025 at the Department of Neurosurgery, Qilu Hospital. The primary outcome was the change in motor function, including the Burke-Fahn-Marsden Dystonia Rating Scale movement (BFMDRS-M) and disability subscale (BFMDRS-D) at 3 days before DBS (baseline) surgery and 1, 3, 6, and 12 months after surgery. Secondary outcomes included health-related quality of life, sleep quality status, depression severity, and anxiety severity at 3 days before and 12 months after DBS surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Primary Meige syndrome was diagnosed by an experienced neurologist.
2. All patients had received systematic and regular treatment for at least 1 year before surgery, including oral drugs and local injection of botulinum toxin A, but the efficacy was not apparent, as the ability to engage with daily life and the quality of life of the patients significantly decreased.
3. Tere were no other serious systemic diseases, such as severe organic heart disease, severe lung, liver and kidney dysfunction, and coagulation dysfunction.
4. Tere was no history of neurological diseases other than Meige syndrome, such as Parkinson's disease or severe cognitive dysfunction.
5. Tere were no serious psychiatric disorders, such as schizophrenia.
6. Preoperative head magnetic resonance imaging (MRI) examinations were normal. Patients of missing follow-up and incomplete clinical data were excluded from the cases.

Exclusion Criteria:

1. Unilateral facial spas and blepharospasm.
2. Patients with severe disease such as coronary heart disease, stroke.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in motor function | 12 months after DBS
  The primary outcome was the change in motor function, including the Burke-Fahn-Marsden Dystonia Rating Scale movement (BFMDRS-M)at 3 days before DBS (baseline) surgery and 1, 3, 6, and 12 months after surgery.

SECONDARY OUTCOMES:
health-related quality of life | 12 months after DBS
  Secondary outcomes included health-related quality of life (EuroQol Five Dimensions Questionnaire) at 3 days before and 12 months after DBS surgery.
sleep quality status | 12 months after DBS
  Secondary outcomes included sleep quality status (Pittsburgh Sleep Quality Index) at 3 days before and 12 months after DBS surgery.
Mental syndrome | 12 months after DBS
  Secondary outcomes included depression severity, and anxiety severity including Hamilton Depression Scale (HAMD) scores at 3 days before and 12 months after DBS surgery.
Mental syndrome | 12 months after DBS
  Secondary outcomes included depression severity, and anxiety severity including Hamilton Anxiety Scale (HAMA) scores at 3 days before and 12 months after DBS surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Chao Zhang, Jinan, Shandong, China